CLINICAL TRIAL: NCT04332341
Title: A Pilot Study of Nicotinamide Riboside Supplementation in Allogeneic Hematopoietic Cell Transplantation
Brief Title: Study of Nicotinamide Riboside Supplementation in Allogeneic Hematopoietic Cell Transplantation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2Z20
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Allogeneic Hematopoietic Cell Transplantation
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nicotinamide riboside (NR) (Experimental)
  Interventions: Drug: Nicotinamide riboside (NR)

INTERVENTIONS:
Drug: Nicotinamide riboside (NR) — Nicotinamide riboside, PO, 500mgtwice daily for 21, 28, and 35 days

SUMMARY:
The purpose of this study is to find a safe and tolerable way to improve engraftment after transplant. Research studies have shown that adding nicotinamide riboside to donor cells has the potential to increase blood stem cell numbers and potentially decrease the time to engraftment. Also, nicotinamide riboside, TRU NIAGEN (the study drug) is a type of vitamin B supplement that the general public can get without a prescription and is well tolerated.

DETAILED DESCRIPTION:
This is a single-center, pilot feasibility study of NR supplementation in allogeneic (donor) HCT in which the study team is seeking to obtain preliminary data on any beneficial effect of increasing NAD+ levels in-vivo to facilitate engraftment. Engraftment is defined as the process during which transplanted stem cells begin to grow in the bone marrow and produce new white blood cells, red blood cells, and platelets. It takes about 14 to 24 days for donor cells to engraft after infusion, and the time between which blood counts fall to the time when they recover is a very critical period. Transfusions are frequently required to prevent bleeding and antibiotics are needed to prevent infections during this critical time period. Shortening the time of engraftment decreases these risks and can improve long-term health status.

The primary objectives of this study is to evaluate safety and tolerability of NR supplementation

The secondary objective of this study is to evaluate neutrophil and platelet recovery after HCT

ELIGIBILITY:
Inclusion Criteria:

* All disease indications for allogeneic hematopoietic cell transplantation except for myelofibrosis.
* Subject must meet program eligibility criteria* for myeloablative conditioning alloHCT and plan to undergo myeloablative conditioning.
* HLA-identical related donor or unrelated human donor source with bone marrow graft.
* Subjects must provide a written informed consent.

Exclusion Criteria:

* History of allergy or intolerance to NR precursor compounds, including niacin or nicotinamide
* Pregnant or breastfeeding women are excluded from this study since allogeneic HCT is a strict contraindication.
* Subjects with uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-19 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent of participants who receive >75% of scheduled doses. | day +7
  Tolerability of NR in allogeneic HCT recipients, defined as 8 or more of 15 participants (i.e. at least 50% of enrolled subjects) able to receive >75% of their scheduled doses (overall rate 53%, 95% confidence intervals 33%-86%). This will include both patients who discontinue NR due to study drug related toxicity and patients who are not able to stay on NR due to transplant related toxicity that limits ability to take the drug
Percent of participants who receive >75% of scheduled doses. | day +14
  Tolerability of NR in allogeneic HCT recipients, defined as 8 or more of 15 participants (i.e. at least 50% of enrolled subjects) able to receive >75% of their scheduled doses (overall rate 53%, 95% confidence intervals 33%-86%). This will include both patients who discontinue NR due to study drug related toxicity and patients who are not able to stay on NR due to transplant related toxicity that limits ability to take the drug
Percent of participants who receive >75% of scheduled doses. | day +21
  Tolerability of NR in allogeneic HCT recipients, defined as 8 or more of 15 participants (i.e. at least 50% of enrolled subjects) able to receive >75% of their scheduled doses (overall rate 53%, 95% confidence intervals 33%-86%). This will include both patients who discontinue NR due to study drug related toxicity and patients who are not able to stay on NR due to transplant related toxicity that limits ability to take the drug
Percent of participants experiencing a CTCAE 5.0 grade 3 or higher related to the study drug | day +7
  Safety of NR in allogeneic HCT recipients as measured by percent of participants experiencing a CTCAE 5.0 grade 3 or higher that is related to the study drug
Percent of participants experiencing a CTCAE 5.0 grade 3 or higher related to the study drug | day +14
  Safety of NR in allogeneic HCT recipients as measured by percent of participants experiencing a CTCAE 5.0 grade 3 or higher that is related to the study drug
Percent of participants experiencing a CTCAE 5.0 grade 3 or higher related to the study drug | day +21
  Safety of NR in allogeneic HCT recipients as measured by percent of participants experiencing a CTCAE 5.0 grade 3 or higher that is related to the study drug

SECONDARY OUTCOMES:
Median days to neutrophil recovery after HCT | Up to 100 days from start of treatment
  Median and range of days to neutrophil recovery after HCT. Recovery defined as first day of three consecutive days with absolute neutrophil count 500 cells/mm3 (0.5 x 109/L) or greater
Median days to platelet recovery after HCT | Up to 100 days from start of treatment
  Median and range of days to Platelet recovery after HCT. Recovery defined as first day of three consecutive days with platelet count 20,000/mm3 (20 x 109/L) or greater and unsupported by platelet transfusions.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Sobecks, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared publicly